CLINICAL TRIAL: NCT06780917
Title: Validating the On-line Creyos Cognitive Assessment Platform in Older Adults With Major Depressive Disorder or Mild Cognitive Impairment
Acronym: Creyos-MD
Status: Recruiting | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Krembil Foundation (Unknown)
Responsible Party: Principal Investigator, Benoit Mulsant, Professor, Labatt Family Chair, Department of Psychiatry, University of Toronto; Senior Scientist, Centre for Addiction and Mental Health, Centre for Addiction and Mental Health
Other Study IDs: 4912
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment (MCI); Major Depressive Disorder, Remitted; Healthy Controls Group - Age and Sex-matched
Keywords: Neuropsychological testing; Mild Cognitive Impairment; Online neuropsychological testing; Cognition
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MCI: Individuals diagnosed with Mild Cognitive Impairment
- Major Depressive Disorder in remission: Individuals with major depressive disorder in remission, with no active symptoms of depression
- Control participants: Individuals with no history of psychiatric illness, not currently taking any psychotropic medications

SUMMARY:
The goal of this observational study is to validate the Creyos online cognitive assessment platform in individuals with mild cognitive impairment, or remitted major depressive disorder. The main objectives of this research are:

1. To confirm the feasibility of administering the Creyos cognitive battery to older adults with Mild Cognitive Impairment MCI) or Major Depressive Disorder in remission (rMDD).
2. To determine whether the Creyos battery can detect changes in cognition that are predictive of changes on paper-and-pencil neuropsychological testing ("gold standard") over up to five years.

Participants will complete both in-person neuropsychological testing yearly as well as the Creyos online battery quarterly for up to 5 years, to allow us to compare performance on these two batteries over time.

ELIGIBILITY:
General Inclusion Criteria:

* Ability to read and communicate in English
* Availability of a study partner who has regular contact with the participant

General Exclusion Criteria:

* Lifetime DSM 5 diagnosis of schizophrenia, bipolar disorder, or OCD
* DSM 5 diagnosis of alcohol or other substance use disorder within the past 12 months
* High risk for suicide
* Significant neurological conditions (e.g. stroke, seizure disorder, MS)
* Unstable medical illnesses (e.g. uncontrolled diabetes mellitus or hypertension)
* Taking anticonvulsants or other psychotropic medication that may interfere with cognitive testing that cannot be safely tapered and discontinued
* Current depressive symptoms defined as a MADRS score of 10 or above

Specific Eligibility Criteria for the MCI Group:

Inclusion:

* Aged 60 or older
* Meets DSM 5 criteria for Minor Neurocognitive Disorder ("MCI")

Exclusion:

* Having taken a cognitive enhancer within the past 6 weeks

Specific Eligibility Criteria for the rMDD Group:

Inclusion:

* Aged 65 or older
* Meets DSM 5 criteria for one or more major depressive episode(s) (MDE) during their adult life (i.e. 18 years of age or older) with: (a) an offset of 2 months to 5 years from the screening visit date, or (b) an offset of 5 years or more, with at least one MDE receiving medical attention (e.g. previously been on an antidepressant, saw a psychiatrist, primary care physician, or had a previous hospitalization

Exclusion:

* Having taken a cognitive enhancer within the past 6 weeks
* Having received electroconvulsive therapy (ECT) within 6 months of baseline neuropsychological testing

Specific Eligibility Criteria for the Control Group:

Inclusion:

* Aged 60 or older

Exclusion:

* Meets DSM 5 criteria for MDD at anytime during their lifetime
* Meets DSM 5 criteria for Minor Neurocognitive Disorder ("MCI")

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit participants with MCI, rMDD or controls in Toronto, Ontario, Canada who are available to come to the Centre for Addiction and Mental Health once per year for up to 5 years for in-person assessments
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Creyos Battery Administration | Upon completion of the Creyos online cognitive platform, approximately every three months, for up to 5 years
  To determine the feasibility of administering the Creyos online cognitive platform in individuals with MCI and major depressive disorder in remission, participants will complete two questionnaires after every completion of the Creyos battery. Participants will be asked to complete the System Usability Scale (10 items). Scores on the System Usability Scale range from 0 to 100, with higher scores indicating greater usability. We will look at the total score to determine how easy the participants find the Creyos online cognitive platform to use, and if usability increases with exposure to the platform.
Feasibility of the Creyos Battery | Upon completion of the Creyos online cognitive platform, approximately every three months, for up to 5 years
  To determine the feasibility of administering the Creyos online cognitive platform in individuals with MCI and major depressive disorder in remission, participants will complete two questionnaires after every completion of the Creyos battery. Participants will be asked to complete the User Burden Scale (20 items). Scores on the User Burden Scale range from 0 to 80, with higher scores indicating greater user burden. We will look at the total score to determine how easy the participants find the Creyos online cognitive platform to use, and if usability increases with exposure to the platform.
Validity of the Creyos Platform | In-person testing is completed yearly, and the Creyos online battery is complete quarterly, for up to 5 years
  To determine the validity of the Creyos online platform, we will compare the single test scores, domain composite scores and global composite scores between the in-person paper-and-pencil neuropsychological tests ("gold standard") and the Creyos online battery.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided